CLINICAL TRIAL: NCT02033876
Title: Effect of Delayed-Release Ursodeoxycholic Acid on Insulin Sensitivity, Gastric Emptying and Body Weight in Overweight or Obese Patients With Type 2 Diabetes on Metformin Treatment
Brief Title: Ursodiol on Insulin Sensitivity, Gastric Emptying and Body Weight With Type 2 Diabetes on Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Professor of Medicine, Pharmacology and Physiology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-004908
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ursodiol (Experimental): Ursodeoxycholic acid (UDCA) 600mg in delayed (ileocolonic)-release to be taken twice daily
  Interventions: Drug: Ursodiol
- Placebo (Placebo Comparator): matching placebo capsules to be taken twice daily
  Interventions: Drug: Ursodiol

INTERVENTIONS:
Drug: Ursodiol
  Other Names: Ursodeoxycholic acid

SUMMARY:
This study will evaluate whether bile acids are able to increase insulin sensitivity and enhance glycemic control in T2DM patients, as well as exploring the mechanisms that enhance glycemic control. These observations will provide the preliminary data for proposing future therapeutic as well as further mechanistic studies of the role of bile acids in the control of glycemia in T2DM.

DETAILED DESCRIPTION:
Background: Intra-jejunal administration of bile acids improves insulin sensitivity.

Hypothesis: The bile acid, ursodeoxycholic acid (UDCA) in delayed (ileocolonic)-release formulation, stimulates bile acid membrane receptor (TGR-5) and farnesol X (FXR) receptors in the ileum and colon, increasing the secretion of Fibroblast growth factor 19 (FGF-19), GLP-1, oxyntomodulin (OXM), and Peptide (PYY3-36), improving insulin sensitivity and inducing weight loss.

Aim: To study the effect of an ileocolonic formulation of UDCA on insulin sensitivity, postprandial plasma glycemia and incretin levels, gastric emptying and body weight in overweight or obese type 2 diabetic subjects on monotherapy with metformin.

Study design: This is a single center, placebo-controlled, parallel group, single dose randomized controlled trial to study the effect of delayed (ileocolonic)-release UDCA 600 mg twice daily on insulin sensitivity, gastric emptying of liquids and solids (measured by scintigraphy)and weight loss in overweight or obese type 2 diabetic subjects. Participants will be receiving monotherapy with metformin. Blood samples will be collected at defined times to measure glycemia and the incretin (GLP-1, OXM, PYY3-36) fasting levels and responses to the meal.

Anticipated Results: In comparison with placebo, UDCA will increase insulin sensitivity, enhance glycemic control, increase postprandial incretins, and delay gastric emptying (GE) of liquids.

Significance: This study will prove that ileocolonic-release UDCA enhances glycemic control in T2DM patients.

ELIGIBILITY:
Overweight or Obese subjects with BMI> 25 Kg/m2 with Type 2 Diabetes mellitus on Metformin, receiving standard of care for Type 2 DM. Otherwise individuals who are not currently on treatment for cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, endocrine (other than T2DM) and unstable psychiatric disease.

Men or women. Women of childbearing potential will have a negative pregnancy test before initiation of medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Calderon G, McRae A, Rievaj J, Davis J, Zandvakili I, Linker-Nord S, Burton D, Roberts G, Reimann F, Gedulin B, Vella A, LaRusso NF, Camilleri M, Gribble FM, Acosta A. Ileo-colonic delivery of conjugated bile acids improves glucose homeostasis via colonic GLP-1-producing enteroendocrine cells in human obesity and diabetes. EBioMedicine. 2020 May;55:102759. doi: 10.1016/j.ebiom.2020.102759. Epub 2020 Apr 25. PMID 32344198
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Ursodiol: Ursodeoxycholic acid (UDCA) 600mg in delayed (ileocolonic)-release to be taken twice daily
  Ursodiol
- Placebo: matching placebo capsules to be taken twice daily
  Ursodiol
Period: Overall Study
Arm/Group | Ursodiol | Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ursodiol | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62.5 [59 to 64] | 57 [47.5 to 64] | 58.9 [47.5 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Area Above Basal (AAB) for Glucose
Description: Mixed meal glucose results are used to calculate the area above basal (AAB) for glucose. The glycemic index of a food is defined as the incremental area under the two-hour blood glucose response curve (AUC) following an overnight fast and ingestion of a food with a certain quantity of available carbohydrate (usually 50 g).
Time Frame: baseline, post-treatment approximately 14 - 17 days
Measure: Median (Inter-Quartile Range); unit: mg/dL x min
Arm/Group | Ursodiol | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL x min | 66458 [53501 to 75478] | 72566 [55654 to 93006]
Statistical Analysis 1: Comparison: Ursodiol vs Placebo; Test type: Superiority; p = 0.43, ANCOVA

2. Secondary Outcome: Change in Fasting Glucose
Description: Serum glucose measurements taken after 10 hours of fasting.
Time Frame: baseline, post-treatment approximately 14 - 17 days
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Ursodiol | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL | 142 [125.7 to 158.8] | 155.7 [126.8 to 166.2]
Statistical Analysis 1: Comparison: Ursodiol vs Placebo; Test type: Superiority; p = 0.65, ANCOVA

3. Secondary Outcome: Change in Insulin Sensitivity
Description: Insulin sensitivity will be calculated by the oral minimal model.
Time Frame: baseline, post-treatment approximately 14 - 17 days
Measure: Median (Inter-Quartile Range); unit: mg/dL x minutes
Arm/Group | Ursodiol | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL x minutes | 19983 [15260 to 28298] | 19086 [13952 to 24038]

4. Secondary Outcome: Gastric Emptying of Liquids (T1/2)
Description: The time for half of the ingested liquids to leave the stomach. Following a meal with milk labeled with indium In111 diethylenetriaminepentaacetate (0.1 mCi), gastric emptying of liquids was assessed with scintigraphy imaging.
Time Frame: post-treatment, approximately 14-17 days
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Ursodiol | Placebo
Number analyzed (Participants) | 12 | 12
minutes | 63.2 [50 to 78.1] | 63.6 [50 to 73.8]
Statistical Analysis 1: Comparison: Ursodiol vs Placebo; Test type: Superiority; p = 0.37, ANCOVA

5. Secondary Outcome: Gastric Emptying of Solids (T1/2)
Description: The time for half of the ingested solids to leave the stomach. Following a meal consisting of two eggs labeled with technetium Tc 99m sulfur colloid (1 mCi) served with 50g of Canadian bacon and one slice of bread gastric emptying of solids was assessed with scintigraphy imaging.
Time Frame: post-treatment, approximately 14-17 days
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Ursodiol | Placebo
Number analyzed (Participants) | 12 | 12
minutes | 167.5 [142.7 to 215.4] | 172.3 [135.3 to 180.9]
Statistical Analysis 1: Comparison: Ursodiol vs Placebo; Test type: Superiority; p = 0.51, ANCOVA

6. Secondary Outcome: Change in Weight
Description: Change in subject's weight, in kilograms
Time Frame: baseline, post-treatment approximately 14 - 17 days
Measure: Median (Inter-Quartile Range); unit: kilograms
Arm/Group | Ursodiol | Placebo
Number analyzed (Participants) | 12 | 12
kilograms | 93.6 [85.7 to 105.4] | 101.9 [85.6 to 114.8]
Statistical Analysis 1: Comparison: Ursodiol vs Placebo; Test type: Superiority; p = 0.4, ANCOVA

7. Secondary Outcome: Change in Body Mass Index
Description: Change in subjects BMI, in kilograms per meter squared.
Time Frame: baseline, post-treatment approximately 14 - 17 days
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | Ursodiol | Placebo
Number analyzed (Participants) | 12 | 12
kg/m^2 | 33.1 [29 to 38.5] | 32.3 [30.1 to 37.3]
Statistical Analysis 1: Comparison: Ursodiol vs Placebo; Test type: Superiority; p = 0.8, ANCOVA

8. Secondary Outcome: Change in FGF-19
Description: Change in fasting fibroblast growth factor (FGF)-19 expression.
Time Frame: baseline, post-treatment approximately 14 - 17 days
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Ursodiol | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL | 52.2 [33.8 to 100] | 90.2 [56.8 to 143.5]
Statistical Analysis 1: Comparison: Ursodiol vs Placebo; Test type: Superiority; p = 0.006, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the subject's participation in the study, approximately five weeks.
Arm/Group | Ursodiol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes